CLINICAL TRIAL: NCT07155213
Title: Feasibility of Vigorous Extended Reality Exergaming on Cardiometabolic Health in Youth With Mobility Disabilities: A Case Series
Brief Title: Adapted High-Intensity Virtual Reality Exergaming
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Byron Lai, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300014468
Record Dates: First submitted 2025-08-12; First posted 2025-09-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cerebral Palsy
Keywords: active video gaming; telehealth; telerehabilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: Virtual reality high-intensity exercise in either the seated or standing position.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Exergaming Intervention (Experimental): High-intensity active video gaming at the home.
  Interventions: Behavioral: Virtual reality exergaming

INTERVENTIONS:
Behavioral: Virtual reality exergaming — High-intensity active video gaming using head-mounted display.

SUMMARY:
This study will test the acceptability and benefits of a home-based high-intensity virtual reality exercise program for young people with physical disabilities. The program will last 6 weeks. There will be a total of two visits to the laboratory for exercise-related health assessments. The program includes head-mounted displays (Meta Quest) and off-the-shelf games.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese (based on CDC body mass index normative ranges for age and sex)
* physically inactive (<150 min/week of moderate exercise)
* Gross Motor Function Classification System level (GMFCS) levels I-IV
* Physician clearance to participate
* Wifi internet access at home

Exclusion Criteria:

* Complete blindness or deafness
* GMFCS level V
* Unable to communicate in English
* Prone to photosensitive seizures
* Pregnant (due to radiation from a Dual Energy X-ray Absorptiometry [DXA] scan

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Total lean mass | week 0, week 7
  lbs
Total fat mass | Week 0, Week 7
  lbs
Systolic blood pressure | Week 0, week 7
  mmHg
high sensitivity C-reactive protein (hsCRP) | Week 0, Week 7
  mg/L
hemoglobin A1c (HbA1C) | Week 0, week 7
  mmol/mol
fasting insulin | Week 0, week 7
  μIU/mL
Total cholesterol | Week 0, week 7
  mg/dL
Low-density lipoprotein | Week 0, week 7
  mg/dL
High-density lipoprotein | Week 0, week 7
  mg/dL
Diastolic blood pressure | Week 0, week 7
  mmHg

SECONDARY OUTCOMES:
Peak oxygen consumption (pVO2) | Week 0, Week 7
  mlkg/min
Total work output | Week 0, Week 7
  watts
Resting heart rate | Week 0, week 7
  beats/min

OTHER OUTCOMES:
Adolescent Food Habits Checklist | Week 0, week 7
  The short survey includes 23 items where the person can respond with True and False to a variety of healthy eating habit questions. The survey is scored by a frequency count of 1 point for each 'healthy' response. Final score achieved by summing number of 'healthy' responses x (23 / number of items completed).
Total minutes of intervention exercise | Week 0 - Week 6
  Total minutes of virtual reality exercise performed each week will be recorded and divided by the total prescribed 240 minutes per week across the 6 week program.
Total vigorous-intensity minutes of intervention exercise | Week 0 - Week 6
  Vigorous-intensity minutes of virtual reality exercise performed each week will be recorded and divided by the target of 187 minutes per week across the 6 week program. Vigorous-intensity will be defined as >75% of age predicted heart rate maximum.
Frequency of technical problems with the technology and exercise | Week 0 - 7
  Participant report: 1) frequency of problems reported
Type of technical problems with the technology and exercise | Week 0 - 7
  Participant report: 1) Type of problem

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Wellness Health and Research Facility, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
All raw data will be published.